CLINICAL TRIAL: NCT05770336
Title: STUDIO DELLE MANIFESTAZIONI CARDIOVASCOLARI A LUNGO TERMINE MEDIANTE TECNICHE DI IMAGING
Acronym: LONG-COVID
Status: Completed | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Collaborators: Rete cardiologica IRCCS (Unknown)
Responsible Party: Principal Investigator, Agricola Eustachio, PI, IRCCS San Raffaele
Other Study IDs: LONG-COVID
Record Dates: First submitted 2023-03-12; First posted 2023-03-15 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Cardiac Complication; COVID-19 Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with previous hospitalization for Covid-19 infection

SUMMARY:
The aim of the project is to identify the prevalence and characteristics of long-term cardiovascular changes in Covid-19 infection.

DETAILED DESCRIPTION:
In the follow-up of patients with Covid-19 infection, persistence of cardiovascular symptoms is common. Studies of the acute phase of Covid-19 infection have shown a significant prevalence of acute myocardial damage (15-44%), and imaging studies have confirmed the presence of structural changes in the pericardium and myocardium several months after the acute phase.

The aim of the project is to identify the prevalence and characteristics of long-term cardiovascular changes in Covid-19 infection.

The study is a continuation of the project "Registry "CARDICoVRISK"" which collected data on cardiovascular changes during the acute phase and shortly after the acute phase. The study design is retrospective observational. The study plans to enroll 240 patients hospitalized during the acute phase of COVID-19 infection. Patients will be collected at three separate centers. Enrolled patients will undergo a baseline evaluation by history, physical examination, laboratory tests, ECG, 6-minute walking test and echocardiogram.

If alterations in left ventricular or right ventricular systolic function are found, as per the standard clinical approach, a cardiac MRI examination will be evaluated.

Identification of patients with cardiac changes is of paramount importance as they may benefit from early initiation of cardioprotective therapy and may need different follow-up strategies.

ELIGIBILITY:
Inclusion Criteria:

* Patient with previous hospitalization for Covid-19 infection confirmed by pharyngeal molecular swab
* Adult patients between 18 and 90 years of age
* Signature of informed consent

Exclusion Criteria:

* Patient with poor echocardiographic acoustic window impairing the performance of the examination
* Patients with atrial fibrillation
* Patients with ischemic or nonischemic heart disease with known decreased left ventricular systolic function

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with previous hospitalization for Covid-19 infection
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2022-03-09 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Identify the long-term myocardial damage and compare it with the prevalence and extent of acute myocardial damage. | 9 months
  The main purpose of this study is to identify the long-term myocardial damage and compare it with the prevalence and extent of acute myocardial damage. The anatomical and functional substrates of cardiovascular manifestations will be analyzed by basic and advanced echocardiographic technologies

CONTACTS AND LOCATIONS:
Overall Officials: Eustachio Agricola, MD, Study Director — IRCCS San Raffaele
Locations (1):
- IRCSS San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided